CLINICAL TRIAL: NCT05568849
Title: Optical Coherence Tomography Angiography (OCTA) to Assess Cardiac Output and Cerebral Perfusion at the Time of Children's Cardiac Surgery
Brief Title: Optical Coherence Tomography Angiography (OCTA) in Children's Cardiac Surgery
Acronym: OCTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21HL23; 314744 (Version 2.0) (Other: IRAS)
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Congenital Heart Disease; Children, Only
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCTA measurement arm (Experimental): There is only one arm in the study and patient care will not be changed. Additional measurements will be obtained over and above usual patient care in the OCTA measurement arm as detailed in the protocol.
  Interventions: Diagnostic Test: OCTA measurements

INTERVENTIONS:
Diagnostic Test: OCTA measurements — OCTA images will be obtained from the retina at 1-3 time points around the time of children's heart surgery

SUMMARY:
Around 3500 children including 1,000 babies a year in the UK require heart surgery. Open-heart repairs involve the heart being stopped, while blood is pumped around the body using a cardiopulmonary bypass machine. Following complex operations, the patient may temporarily develop poor heart function, leading to reduced organ blood supply. Low heart output leads to post-operative complications or even death. The current methods to assess cardiac output and to see if vital organs, especially the brain, are receiving enough blood flow, are indirect and can be inaccurate. If we find a better way to detect and then avert or ameliorate periods of poor cardiac output and / or reduced brain perfusion, then this would be helpful for clinicians and could lead to better outcomes for children.

We believe that optical coherence tomography angiography (OCTA), a non-invasive way to image the blood vessels in the retina at the back of the eye, could help us to assess cardiac output and brain perfusion. The OCTA machine was approved for use in humans in 2019 and given a CE Marking, but it has previously been used mainly in the management of eye diseases. There is a small amount of experience with its use in critically ill adults. We plan a pilot study to see if it is possible to use the OCTA machine at key time points, before, during and after children's heart operations, in 30 patients. We will study the images taken with OCTA machine to see if they are of good quality and we will analyze the images to see whether or not the expected changes in cardiac output and brain perfusion that occur with heart surgery can be detected as changes in blood flow in the back of the eye. Depending on the success of this pilot, we will plan further studies.

DETAILED DESCRIPTION:
• OBJECTIVES

1. To undertake a pilot study in young children undergoing cardiothoracic surgery to treat congenital heart disease involving cardiopulmonary bypass (CPB) at Great Ormond Street Hospital for Children (GOSH) in which OCTA images will be collected.
2. To evaluate any practical barriers to acquiring OCTA images from children around the time of their heart surgery at GOSH, ensuring that the conduct of the anaesthetic and surgery are not disturbed.
3. To process and review de identified OCTA images to see whether or not they provide potentially meaningful clinical data about peri-operative changes in cardiac output and cerebral perfusion for children undergoing surgery with CPB.

   • HYPOTHESES

<!-- -->

1. It is feasible to use OCTA to obtain images that can be used to examine regional neuronal microcirculation and better understand peri-operative cerebral blood flow at stages before, during and immediately after cardiopulmonary bypass.
2. There will be detectable, reproducible changes in OCTA readings at different states; pre-CPB, during and post-CPB and that these changes will be reflective of cerebral blood flow at these times.

   A future hypothesis that will not be tested in this pilot study, but could be tested in a later evaluation study:

   OCTA monitoring peri-operatively may lead to better, earlier diagnosis of reduced cardiac output and of impairments to the cerebral circulation in the peri-operative period related to surgery for CHD. This will then enable better individualized approaches to CPB strategy and postoperative care, with potential for patient benefit.

   • RECRUITMENT

   Participants for inclusion in the study will be identified in advance by reviewing the list of patients scheduled for cardiac surgery requiring cardiopulmonary bypass available from the cardiac theatre coordinator. Their eligibility will be confirmed by the absence of exclusion criteria and ensuring the participant meets all inclusion criteria.

   When the patient and parent(s) attend their pre-cardiac surgical assessment clinic, they will be given a patient information leaflet and if they express interest, they will be given an opportunity to discuss participation in the study. If a child is an inpatient prior to surgery then this will occur on the cardiology ward. Informed consent will be taken either in the pre-cardiac surgical assessment day case unit or the cardiology ward.

   • RESEARCH SUBJECT CONFIDENTIALITY

   Patient confidentiality will be of utmost importance during data collection, and we will make every effort to protect the privacy of each research subject. We will not collect nor hold patient identifiers and we will collect the minimum clinically important information about each patient necessary to complete the study objectives.
   * DRUG INFORMATION

   The research entails the administration of a licensed medication for the purposes of the research, and not for clinical benefit. The licensed medication is eye drops, of a type that are licensed for use in this age group and are routinely used to examine the back of the eye (the fundus of the eye) by eye specialists.

   I) TROPICAMIDE

   The study will use Minims tropicamide drops (Bausch & Lomb UK Limited); a topical mydriatic and cycloplegic agent used to dilate the pupil and temporarily paralyse the lens 20 minutes before eye examination. This is needed so that the images of the fundus of the eye can be obtained. The duration of effect is 60-90 minutes and up to 6 hours. We will only examine one of the two eyes and will make the clinical care team fully aware of which eye we are studying.

   DOSE - We will use the standard clinical paediatric dosing regimen per the British National Formulary for Children.

   II) PHENYLEPHRINE EYE DROPS

   Drug information Minimis Phenylephrine Hydrochloride 2.5% w/v eye drops. DOSE -We will use the standard clinical paediatric dosing regimen per the British National Formulary for Children.

   • OCTA EQUIPMENT

   The study entails the use of a CE marked device which has been used extensively to image the eyes of children and adults, but not in the setting of paediatric cardiac surgery.

   • DATA PROCESSING AND STORAGE

   OCTA images and other pseudonymized study data will be stored with patient study ID only and no identifying information.

   Images will be reviewed for quality. Images at different time points will be reviewed for evidence of change. Study data will be held for up to three years after the end of the study.

   • FOLLOW-UP

   Patients and their families will be contacted when they are in the ward and the child has recovered, just before they are discharged from hospital for a brief follow-up interview about any post-procedure adverse events or feedback about participation. At this time, we will ask the parent and the child for feedback about participating in the research. We will ask whether or not they have noticed any visual symptoms or eye irritation.

   • STATISTICS

   We anticipate that in our initial studies we may generate images of inferior quality and as such we need a sufficient sample size to accommodate a 'learning curve'.

   Image quality analysis - this metric is an integer between 1 and 200 provided by the OCTA machine internal software, which will be grouped as poor, medium or good based on the OCTA software.

   Vessel density is a % between 0-100, again provided by the OCTA internal software, the vessel density at the study timepoints will be used to look for evidence of change.

   Once we have learned how to acquire clinically usable images within the setting of children's heart surgery, we will then set out to compare images at the three time points to look for evidence of change. We have included a sample size of 30 as a reasonable number likely to see us through a learning phase through to providing sufficient good quality images for at least two time points such that we can detect a change of at least 15% flow reduction from pre-operative time point and the later time points.

   • ADVERSE EVENT REPORTING

   The primary investigators accept responsibility of reporting adverse events by completing an Adverse Event (AE) form including information on the seriousness of the adverse event, assessing whether or not it is a direct consequence of the research study and proposing any further action. The primary investigators are aware of and accept the responsibility of the adverse event reporting requirements of investigators as well as timelines for reporting as defined in the Research Ethics Board Adverse Event Reporting Requirements.

   All serious, unexpected adverse drug reactions to the study medication will be reported to the MHRA through the Yellow Card Scheme within 15 calendar days or for death or life-threatening events, within 7 calendar days. In the latter case, a follow-up report must be filed within 8 calendar days.

   • DATA SAFETY MONITORING

   The Data Safety Monitoring Board (DSMB) will be responsible for oversight of data and safety. The DSMB for this study will be chaired by Mr Nigel Drury Cardiothoracic Surgeon and Clinical Trials expert Birmingham Children's Hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery for congenital heart disease including both repair and palliation involving CPB.
* Patients under 10 years of age.

Exclusion criteria

* Patients undergoing emergency or salvage surgery.
* Patients who are clinically unstable prior to the operation.
* Patients with known hypersensitivity to tropicamide drops or to any ingredient in its formulation.
* Patients with known hypersensitivity to phenylephrine drops or to any ingredient in its formulation.
* Patients with known high intra-ocular pressure or personal or family history of glaucoma.
* Patients who are taking any of the following medications which may interact with phenylephrine eye drops: anti-hypertensive medications, monoamine oxidase inhibitors, tricyclic antidepressants, cardiac glycosides or quinidine.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the feasibility of taking at least two sets of good quality OCTA images per patient during the conduct of cardiac surgery | 1-3 hours
  Feasibility measure

SECONDARY OUTCOMES:
The acceptability of the study procedures to members of the clinical care team based on a Likert rating scale. | 2-3 hours
  acceptability measure
Change in blood flow measured in the retina by OCTA | 1-3 24 hours
  Quantitative change between timepoints 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Brown, MD MPH, Principal Investigator — Great Ormond Street Hospital NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pilot study. If successful pilot will be published subject to peer review.